CLINICAL TRIAL: NCT00004345
Title: Study of Dietary N-3 Fatty Acids in Patients With Retinitis Pigmentosa and Usher Syndrome
Status: Terminated | Type: Observational
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Oregon Health and Science University (Other)
Other Study IDs: 199/11904; OHSU-2650
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2002-07

CONDITIONS: Usher Syndrome; Retinitis Pigmentosa
Keywords: Usher syndrome; ophthalmologic disorders; rare disease; retinitis pigmentosa
MeSH Terms: conditions — Usher Syndromes; Retinitis Pigmentosa; Rare Diseases

SUMMARY:
OBJECTIVES: I. Examine the concentration of docosahexanoic acid (DHA) and other n-3 fatty acids in plasma, erythrocyte, and adipose tissue in patients with various forms of retinitis pigmentosa and Usher syndrome.

II. Determine the synthesis and catabolism of DHA from linolenic acid in these patients.

III. Determine the synthesis, absorption, and catabolism of DHA under different dietary conditions in these patients.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Patients may participate in one or more of the arms of this study.

Arm I (adipose tissue study): Adipose tissue is collected from the buttocks of patients with Usher II retinitis pigmentosa (RP), patients with non-Usher RP, and control subjects. Dietary histories are obtained from all patients and subjects.

Arm II (isotope study): Patients meeting the same criteria as in arm I receive oral D5-labeled linolenic acid and oral D4-labeled linolenic acid that is dissolved in oil and incorporated into foods. Subjects must avoid eating fish and shellfish during the 35 days of the isotope study. Blood samples are collected at 0, 8, 24, and 48 hours, daily on days 3-7, and then on days 10, 18, and 35.

Arm III (flaxseed oil feeding): Patients with all types of RP and control subjects receive flaxseed oil, a form of linolenic acid, for 12 weeks. Subjects may also receive high oleic safflower oil or olive oil as a control fat for 12 weeks. Subjects complete a diet history at the end of each fatty acid supplementation period. All subjects must follow a diet free of seafood and fish oil supplements.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

* Retinitis pigmentosa, including: Usher syndrome (types I and II) Simplex
* The following inheritance patterns eligible: X-linked recessive; Autosomal dominant; Autosomal recessive

Min Age: 0 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 1999-10

CONTACTS AND LOCATIONS:
Overall Officials: William Connor, Study Chair — Oregon Health and Science University
Locations (1):
- Oregon Health Sciences University, Portland, Oregon, United States

REFERENCES:
- [Derived] Schwartz SG, Wang X, Chavis P, Kuriyan AE, Abariga SA. Vitamin A and fish oils for preventing the progression of retinitis pigmentosa. Cochrane Database Syst Rev. 2020 Jun 18;6(6):CD008428. doi: 10.1002/14651858.CD008428.pub3. PMID 32573764